CLINICAL TRIAL: NCT02762747
Title: Pre-peritoneal Drainage Versus No Drainage After Totally Extra-peritoneal Hernioplasty for Inguinal Hernia - a Randomised Controlled Study
Brief Title: Randomised Controlled Trial on Pre-peritoneal Drainage After Totally Extra-peritoneal Hernioplasty for Inguinal Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The University of Hong Kong-Shenzhen Hospital (Other)
Responsible Party: Principal Investigator, Dr. Joe King-Man Fan, Consultant, The University of Hong Kong
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HERN-LAPDRAIN-01
Record Dates: First submitted 2016-05-03; First posted 2016-05-05 (Estimated); Last update posted 2016-05-10 (Estimated); Status verified 2016-05

CONDITIONS: Hernia, Inguinal
Keywords: Hernia, Inguinal; Extraperitoneal Hernioplasty; Drain; Mesh Repair; Laparoscopic
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drain (Experimental): preperitoneal suction drainage after laparoscopic totally extra-peritoneal hernioplasty for inguinal hernia
  Interventions: Procedure: preperitoneal suction drainage
- No-drain (No Intervention): No drainage after laparoscopic totally extra-peritoneal hernioplasty for inguinal hernia

INTERVENTIONS:
Procedure: preperitoneal suction drainage — preperitoneal suction drainage after laparoscopic totally extra-peritoneal hernioplasty for inguinal hernia
  Arms: Drain

SUMMARY:
This is a RCT on drain versus no drain after laparoscopic totally extra-peritoneal hernioplasty. We will assess the difference in seroma formation after surgery in 2 two groups by an independent assessor clinically and radiologist to document the size of seroma after surgery. Other secondary outcomes will be measured including post-operative pain, discomfort, analgesic used, patient satisfaction, recurrence of hernia, wound infection, etc.

DETAILED DESCRIPTION:
Inguinal hernia is a common disease and causes significant morbidity if left untreated. With the advances of laparoscopic approach of extra-peritoneal hernioplasty, it significantly reduces the post-operative pain and lead to a better quality of life with higher acceptance to patients.However, similar to traditional Litchenstein approach, post operative seroma formation is still a common problem encountered after surgery. Numerous method has been described to reduce chance of seroma formation, however, none was proven to be effective except pre-peritoneal drainage. There are currently 2 large retrospective non-randomized cohort study to evaluate the effectiveness of preperitoneal drainage available for reference. We therefore study the feasibility and efficacy of preperitoneal drainage with large scale randomized trial.

Patient fulfill inclusion criteria and consent to surgery and study will be recruited. A standardized pre-peritoneal dissection and mesh placement will be adopted. Immediately before deflation of pre-peritoneal space, randomization will be performed by calling research assistant for study group using computer generated code. Drain will be placed for 23 hours after operation and ultrasonography will be performed immediately after removal of drain. USG will be repeated at post-operative 1 week, 1 month, 3 months, 6 months and 1 year after surgery. For non-drain group, a fake drain will be attach to the skin of the wound to achieve double blinding to patients and assessors. In addition to seroma, patient demographics and secondary outcome including post-operative pain score, discomfort, foreign body sensation, patient satisfaction, infection, recurrence, etc will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and below 80
* Male or female patients
* Unilateral inguinal hernia
* First occurrence hernia
* Consent to laparoscopic hernioplasty for inguinal hernia

Exclusion Criteria:

* Inguino-scrotal hernia
* Recurrent inguinal hernia
* Incarcerated hernia
* Bilateral inguinal hernia
* Bleeding tendency
* On anti-platelet agent or anti-coagulant
* Co-morbidies
* Decline or not consent to surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-05; Primary Completion 2018-05 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Seroma formation after TEP hernioplasty | post-operative day 1
  Seroma will be assessed clinically by independent assessor who is blind to the group assigned and also by qualified radiologist who will perform USG to measure the exact size of seroma formation after TEP
Seroma formation after TEP hernioplasty | post-operative day 7
  Seroma will be assessed clinically by independent assessor who is blind to the group assigned and also by qualified radiologist who will perform USG to measure the exact size of seroma formation after TEP
Seroma formation after TEP hernioplasty | post-operative 1 month
  Seroma will be assessed clinically by independent assessor who is blind to the group assigned and also by qualified radiologist who will perform USG to measure the exact size of seroma formation after TEP
Seroma formation after TEP hernioplasty | post-operative 3 month
  Seroma will be assessed clinically by independent assessor who is blind to the group assigned and also by qualified radiologist who will perform USG to measure the exact size of seroma formation after TEP
Seroma formation after TEP hernioplasty | post-operative 6 month
  Seroma will be assessed clinically by independent assessor who is blind to the group assigned and also by qualified radiologist who will perform USG to measure the exact size of seroma formation after TEP
Seroma formation after TEP hernioplasty | post-operative 1 year
  Seroma will be assessed clinically by independent assessor who is blind to the group assigned and also by qualified radiologist who will perform USG to measure the exact size of seroma formation after TEP

SECONDARY OUTCOMES:
Post-operative pain after TEP hernioplasty | post-operative day 1 to day 7, 1 month, 3 month, 6 month, 1 year
  Post-operative pain after TEP hernioplasty will be assessed by self-evaluated VAS questionnaire during initial 7 days after operation. Then will be asked by independent assessor upon follow-up
Analgesic used after after TEP hernioplasty | post-operative day 1 to day 7, 1 month, 3 month, 6 month, 1 year
  Number of analgesic used after after TEP hernioplasty will be assessed by self-evaluated questionnaire during initial 7 days after operation. Then will be asked by independent assessor upon follow-up
Chronic discomfort after TEP hernioplasty | post-operative 1 month, 3 month, 6 month, 1 year
  Chronic discomfort after TEP hernioplasty will be asked by independent assessor upon follow-up
Hernia recurrence after TEP hernioplasty | post-operative 1 month, 3 month, 6 month, 1 year
  Hernia recurrence after TEP hernioplasty will be assessed by independent assessor upon follow-up
Patient satisfaction after TEP hernioplasty | post-operative 1 month, 3 month, 6 month, 1 year
  Patient satisfaction after TEP hernioplasty will be asked by independent assessor upon follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Joe KM Fan, MBBS,MS,FRCS, Study Chair — The University of Hong Kong
Locations (1):
- Department of Surgery, The University of Hong Kong - Shenzhen Hospital, Shenzhen, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ismail M, Garg M, Rajagopal M, Garg P. Impact of closed-suction drain in preperitoneal space on the incidence of seroma formation after laparoscopic total extraperitoneal inguinal hernia repair. Surg Laparosc Endosc Percutan Tech. 2009 Jun;19(3):263-6. doi: 10.1097/SLE.0b013e3181a4d0e1. PMID 19542859
- [Result] Gao D, Wei S, Zhai C, Chen J, Li M, Gu C, Wu H. Clinical research of preperitoneal drainage after endoscopic totally extraperitoneal inguinal hernia repair. Hernia. 2015 Oct;19(5):789-94. doi: 10.1007/s10029-014-1310-0. Epub 2014 Sep 20. PMID 25238803